CLINICAL TRIAL: NCT04361539
Title: Shoulder Muscle Imbalance as a Risk for Shoulder Injury in Elite Adolescent Badminton Players : a Prospective Pilot Study
Brief Title: Shoulder Muscle Imbalance as a Risk for Shoulder Injury in Elite Adolescent Badminton Players
Acronym: BADIRMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: BADIRMS
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2020-04

CONDITIONS: Sport Injury; Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite adolescent badminton players: The population was all the elite adolescent badminton players from a high-level club. We excluded players who had SSI in the 3 months prior to the isokinetic test or had shoulder surgery. They were included and followed from September 2018 to May 2019.

SUMMARY:
Background: To assess the impact of pre-season clinical measures and rotator muscles strength on the risk of significant shoulder injury (SSI) in elite adolescent badminton players Design: Prospective cohort study Participants: Nine elite adolescents badminton players were included and followed from September 2018 to May 2019.

Independent variables: A pre-season visit consisted in clinical and isokinetic shoulder strength testing. Isokinetic internal and external rotator shoulder muscles strength was tested at 60, 120 and 240°/s. Conventional and functional (eccentric-to-concentric) ratios (FR) were calculated. SSI collection was performed by an experienced sport physician.

ELIGIBILITY:
Inclusion Criteria:

* All the elite adolescent badminton players from a high-level club.

Exclusion Criteria:

* Players who had SSI in the 3 months prior to the isokinetic test or had shoulder surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population was all the elite adolescent badminton players from a high-level club
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Isokinetic strength testing (peak torques) at 8 months | Two evaluations, one preseason (september 2018) and one postseason (may 2019) visits
  Shoulder rotator muscles isokinetic strength test, Measures: Peak Torque on internal rotator muscles (IR) and external rotator muscles (ER), in NM (newton.meter)
Change from Baseline Isokinetic strength testing (ratios) at 8 months | Two evaluations, one preseason (september 2018) and one postseason (may 2019) visits
  Shoulder rotator muscles isokinetic strength test, Measures: ratios between external rotator muscles (ER) and internal rotator muscles (IR) (ER:IR), in percent (%)
Clinical measurements, ROM | One evaluation, one preseason visit (september 2018)
  Shoulder internal and external rotation range of motion (ROM)
Clinical measurements TAD | One evaluation, one preseason visit (september 2018)
  table-to-acromion distance (in cm)
Significant Shoulder Injury (SSI) collection (number of injury) | During the badminton season, the number (number, n) of injury was recorded from september 2018 to may 2019
  Significant Shoulder Injury (SSI) collection for the number of injury
Significant Shoulder Injury (SSI) collection (type of injury) | During the badminton season, the type of injury (number, n) was recorded from september 2018 to may 2019
  Significant Shoulder Injury (SSI) collection for the type of injury
Significant Shoulder Injury (SSI) collection (time lost from participation) | During the badminton season, the time lost from participation was recorded (in days) from september 2018 to may 2019
  Significant Shoulder Injury (SSI) collection for time lost from participation due to the injury

CONTACTS AND LOCATIONS:
Overall Officials: Joffrey DRIGNY, MD MSc, Principal Investigator — CHU Caen Normandy
Locations (1):
- CHU Caen Normandie, Caen, France